CLINICAL TRIAL: NCT05954507
Title: Prospective Comparative Multicenter Study Evaluating the Prognostic Interest of PET/MRI in Cardiac Sarcoidosis
Brief Title: Evaluation of the Prognostic Value of PET/MRI in Cardiac Sarcoidosis
Acronym: SARCASTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP191100
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Sarcoidosis
Keywords: Cardiac sarcoidosis; Combined PET/MRI; PET; MRI

STUDY DESIGN:
Intervention Model Description: Prognostic study of a prospective multicenter cohort of patients with suspected cardiac involvement in sarcoidosis.
  All patients with suspected cardiac sarcoidosis meeting the inclusion criteria will be prospectively and consecutively included in each of the study centers. Patients will undergo cardiac PET/MRI within 15 days of inclusion, and will be followed up for 24 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective cohort of patients (Other): Patients with suspected cardiac sarcoidosis
  Interventions: Diagnostic Test: PET/MRI

INTERVENTIONS:
Diagnostic Test: PET/MRI — PET/MRI is a new-generation hybrid camera capable of simultaneously performing FDG positron emission tomography and gadolinium-injected MRI. PET/MRI could be a relevant prognostic marker of progression, and could significantly improve diagnostic performance in patients with suspected cardiac sarcoidosis.

SUMMARY:
Cardiac damage is the second leading cause of death in patients with sarcoidosis, after lung damage. Today's challenge is to diagnose the disease as effectively as possible, and to develop tools for better risk stratification, especially for sudden death, in order to better target therapies and implantable devices, such as corticoids and immunosuppressant.

The hypothesis is that combined PET (Positron Emission Tomography)/MRI (Magnetic Resonance Imaging) could be a relevant prognostic marker of progression, and would significantly improve diagnostic performance in patients with suspected cardiac sarcoidosis (CS). This study will also make it possible to distinguish sequellar fibrosis lesions from granulomatous lesions and assess the therapeutic response. Incorporating PET/MRI into the diagnostic strategy for patients with suspected CS could therefore improve their management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Sarcoidosis defined according to ATS/ERS/WASOG criteria
* Suspicion of cardiac involvement in sarcoidosis:

  * Clinical manifestations (syncope, lipothymia, persistent palpitations, signs of heart failure) and/or
  * Cardiac rhythm or conduction disorder (Mobitz type 2 atrioventricular block (AVB), AVB 3, right or left bundle branch block, Q wave in at least 2 leads, ventricular arrhythmia (ventricular mono/polymorphic complexes> 1000 per 24 h, ventricular tachycardia, ventricular fibrillation), unexplained sustained VT or epsilon wave) and/or
  * Compatible cardiac ultrasound abnormality: left ventricular dilatation, septal thickening or wall thinning (especially basal), segmental kinetic disorder and wall aneurysm without coronary anomaly, altered left ventricular ejection fraction, altered diastolic function, altered right ventricular systolic function.
* Informed patient consent
* Membership of a social security scheme

Exclusion Criteria:

* Psychiatric illness not controlled by treatment
* Claustrophobia
* Known pregnancy or breast-feeding patient
* Unbalanced diabetes (influence on carbohydrate metabolism for PET)
* Previous infarction or known coronary disease
* Known allergy to gadolinium and fluoro-desoxyglucose and their excipients
* Renal insufficiency (Clairance < 30 mL/min/1.73m2)
* Implanted pacemaker not compatible with a 3 Teslas magnetic field
* Patients with ocular metallic foreign bodies, pacemakers, neurostimulators, cochlear implants, metallic heart valves, vascular clips formerly implanted on cranial aneurysms and, in general, any non-removably implanted electronic medical equipment
* Inability or refusal to follow a low-carbohydrate diet for 24 hours, followed by a 6-hour fast required prior to the examination
* Patient unable to hold a 10-second apnea.
* Patient deprived of liberty by judicial or administrative decision
* Patient under legal protection (guardianship, curatorship)
* Participation in other interventional research involving the human person or being in the exclusion period following previous research involving the human person
* Patients under AME

Exclusion criteria (post signature of consent) for women of reproductive age :

- Positive pregnancy test result after inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2030-03-07 (Estimated); Study Completion 2030-03-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a severe cardiological event | Up to 24 months
  Occurrence during follow-up of at least one of the severe cardiological events listed below attributed to sarcoidosis, assessed at 24 months:
  * Death from cardiac causes.
  * Placement of an automatic implantable defibrillator or pacemaker.
  * Conduction disorder (Mobitz type 2 atrioventricular block (AVB), AVB 3, ventricular arrhythmia (ventricular mono/polymorphic complexes > 1000 per 24 h, ventricular tachycardia (VT), ventricular fibrillation), unexplained sustained VT).
  * Degradation of cardiac function of more than 10% of LVEF assessed by transthoracic (TTE) or cardiac MRI.
  * Acute heart failure with no other known cause

SECONDARY OUTCOMES:
Frequency of severe cardiological events between patients with and without Delayde MRI enhancement | Up to 24 months.
  Among patients with hypermetabolic FDG PET uptake
Frequency of severe cardiological events according to each modality of PET/MRI results in terms of Delayde MRI enhancement and hypermetabolic fixation on PET. | Up to month 24.
  MRI- PET-; MRI- PET+; MRI+ PET-; and MRI+ PET+.
Percentage of patients initially well classified (diagnostic accuracy) in terms of probability of cardiac involvement | Up to month 24.
  Percentage of patients initially well classified (diagnostic accuracy) in terms of probability of cardiac involvement (absent, possible, probable or very probable) by each examination (MRI alone, PET alone, or PET/MRI) in relation to the diagnosis established at two years (reference).
Comparison of FDG PET metabolic activity and late gadolinium enhancement of pathological areas before and after treatment. | Up to month 3 and 12.
  For patients with initial pathological MRI-PET.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu MAHEVAS, PHD, Study Director — Assistance public Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION